CLINICAL TRIAL: NCT04226339
Title: Evaluation of Walking Analysis After a Total Knee Arthroplasty With Kinematic Alignment Versus Mechanical Alignment
Acronym: KneeKG Sphere
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0497; 2019-A02288-49 (Other: ANSM)
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Knee Arthroplasty, Total
Keywords: total knee arthroplasty; prosthesis; kinetic alignment; mechanical alignment
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- total knee arthroplasty with a kinetic alignment (Experimental)
  Interventions: Procedure: total knee arthroplasty with a kinetic alignment
- total knee arthroplasty with a mechanical alignment (Active Comparator)
  Interventions: Procedure: total knee arthroplasty with a mechanical alignment

INTERVENTIONS:
Procedure: total knee arthroplasty with a kinetic alignment — During surgery, a SPHERE prosthesis will replace the knee and the femorotibial alignment.
  it will be set to reproduce the preoperative constitutional deformity in varus or valgus as it was measured before surgery
  Arms: total knee arthroplasty with a kinetic alignment
Procedure: total knee arthroplasty with a mechanical alignment — During surgery, a SPHERE prosthesis will replace the knee and the femorotibial alignment.
  It will be set to 180° as defined for a mechanical femorotibial alignment
  Arms: total knee arthroplasty with a mechanical alignment

SUMMARY:
Total knee arthroplasty (TKA) is a treatment for advanced femoro-tibial osteoarthritis. This surgery is justified in case of significant discomfort and failure of medical treatment.

The functional results of TKA are good with a recovery of 6 months - 1 year. Nevertheless, very few patients forget their prostheses. A United Kingdom study assessed patient satisfaction in a cohort of 10,000 patients more than one year after TKA: nearly 20% were not satisfied with their TKA.

The knee is indeed a complex articulation that works differently in the three space plans. Current knee prostheses are trying to replicate this biomechanics and get as close as possible to the anatomy of a native knee.

Bellemans et al. found in 250 asymptomatic patients 32% of men with a constitutional varus greater than 3 ° and 17% of women. Restoration of normal knee function can also be achieved by restoring a moderate constitutional deformity present preoperatively. The objective of the femorotibial alignment was dogmatically fixed at 180° (mechanical femorotibial alignment). In recent years, some surgical teams have attempted to reproduce the preoperative constitutional deformity in varus or valgus with the prosthesis. This femorotibial alignment is called kinematic alignment. This kinematic alignment has already been studied in several randomized studies and has demonstrated improved functional scores. However, these studies focused on specific TKA, which are posterior cruciate TKA, and the assessment was subjective through functional scores. In addition, these TKA were often made with patient specific instrumentation (PSI). Some studies have evaluated walking kinematics after TKA with kinematic alignment. But it was again TKA retaining the posterior cruciate ligament.

The investigators would like to prospectively evaluate the restoration of the medially stabilized TKA walking kinematics (medial-stable TKA or ball in socket stability) implanted with a kinematic alignment compared to a mechanical alignment.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Adults between 55 and 80 years
* Diagnosis of internal or global disabling femorotibial gonarthrosis Indication of total first knee arthroplasty (unilateral), using a Sphere type prosthesis (Medacta)
* Constitutional deformity in varus between 3 ° and 10 °
* Fulfilling the pass conditions of a KneeKG walking test: Unipodal support possible for 1 minute, run for 5 min at a speed of at least 0.8 km / h
* Affiliated to a social security system
* Patients able to understand and fulfill the requirement of the study

Exclusion Criteria:

* TKA bilateral
* TKA to change an Uni-compartmental prosthesis
* History of femoral or tibial fracture
* History of femoral or tibial osteotomy
* Associated gesture at the same time (allograft, osteotomy)
* External femorotibial gonarthrosis
* Angle Hip Knee Ankle > 178 °
* Constitutional distortion> 10 °
* Refusal to participate in the study
* Persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care, persons admitted to a health or social institution for purposes other than research
* Adults subject to a legal protection measure
* breastfeeding or pregnant women
* Patient already participating to another clinical trial that might jeopardize the current trial

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2025-03-07 (Estimated); Study Completion 2029-03-07 (Estimated)

PRIMARY OUTCOMES:
Change of short terms walking speed. | 12 months
  Comparison between the 2 arms, of the walking speed variation between the evaluation before surgery and 1 year after total knee arthroplasty

SECONDARY OUTCOMES:
femorotibial angle in frontal plan | 12 months
  Comparison between the 2 groups of the frontal femorotibial angle measured by the KneeKG system, 12 months after total knee arthroplasty
sagittal femorotibial angle | 12 months
  Comparison between the 2 groups of the sagittal femorotibial angle measured by the KneeKG system, 12 months after total knee arthroplasty
tibia rotation compared to the femur | 12 months
  Comparison between the 2 groups of the tibia rotation angle compared to femur measured by the KneeKG system, 12 months after total knee arthroplasty
maximal knee flexion | 12 months
  Comparison between the 2 groups of the maximal knee flexion measured by the KneeKG system, 12 months after total knee arthroplasty
maximal knee extension | 12 months
  Comparison between the 2 groups of the maximal knee extension measured by the KneeKG system, 12 months after total knee arthroplasty
knee range motion | 12 months
  Comparison between the 2 groups of the knee range motion measured by the KneeKG system, 12 months after total knee arthroplasty
knee functional recovery | 12 months
  Comparison between the 2 groups of the knee functional recovery measured by the International Knee Society (IKS) score 12 months after total knee arthroplasty.
  International Knee Society score : range 0 to 200, a higher score means a better outcome
Ability of the patient to forget his prosthesis | 12 months
  Comparison between the 2 groups of the patient ability to forget his knee prosthesis measured by the Forgotten Joint score (FJS) 12 months after total knee arthroplasty.
  Forgotten Joint Score : range 0 to 100, a higher score means a better outcome
Complications | 12 months
  Comparison between the 2 groups of the proportion of patient with at least one complication including deep infections, prosthesis impairment, knee fracture, surgical revision) during the 12 months after total knee arthroplasty
knee functional recovery | 60 months
  Comparison between the 2 groups of the knee functional recovery measured by the International Knee Society (IKS) score 60 months after total knee arthroplasty.
  International Knee Society score : range 0 to 200, a higher score means a better outcome
Ability of the patient to forget his prosthesis | 60 months
  Comparison between the 2 groups of the patient ability to forget his knee prosthesis measured by the Forgotten Joint score (FJS) score 60 months after total knee arthroplasty.
  Forgotten Joint Score : range 0 to 100, a higher score means a better outcome
Complications | 60 months
  Comparison between the 2 groups of the proportion of patient with at least one complication including deep infections, prosthesis impairment, knee fracture, surgical revision) during the 60 months after total knee arthroplasty

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Lustig, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France